CLINICAL TRIAL: NCT01707836
Title: Genetic Variation and Risk of Pediatric Brain Cancers
Brief Title: Neurofibromatosis Type 1 Brain Tumor Genetic Risk
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201208141
Record Dates: First submitted 2012-10-12; First posted 2012-10-16 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Neurofibromatosis Type 1; Pediatric Brain Tumor
MeSH Terms: conditions — Neurofibromatosis 1

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood or saliva samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Family: Families with a child with Neurofibromatosis Type 1 who has been diagnosed with a brain tumor.

SUMMARY:
This study will analyze DNA samples to determine associations between maternal and offspring genetic factors and pediatric brain tumor development in children with Neurofibromatosis Type 1. Participating families (mother, father, child) will be asked to complete a short questionnaire and provide DNA samples (either saliva or blood). The information gained from your participation may one day help doctors develop strategies to reduce brain tumor risk in individuals with NF1. Please note: there is no therapy associated with this study.

DETAILED DESCRIPTION:
The prenatal period is a developmentally vulnerable time point during which environmental conditions, including nutrition, can have life-long impacts on health.1,2 This is particularly relevant to many childhood cancers that are thought to initiate during pregnancy.3 As a consequence, there has been intense interest in whether prenatal exposures can modulate childhood cancer risk.4-6 It is important to recognize that both maternal and offspring genetic factors including those in nutritional pathways may play an important role in pediatric cancer risk through their effect on the child's exposure to nutrients important in development during the prenatal period. The purpose of this research study is to evaluate whether there are any maternal or offspring genetic factors in the folate pathway that may contribute to the development of brain tumors in children with Neurofibromatosis Type 1 through analysis of DNA samples collected from families.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric participant (born during 1994-2012) with NF1 and diagnosed with a brain tumor
* Biological mother or father (or full sibling if mother or father is unable to participate) able to participate
* All family members (pediatric participant, biological mother, and biological father or full sibling) must be willing to contribute a blood or saliva sample
* ability to understand consent forms

Exclusion Criteria:

-those who do not meet inclusion criteria

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Families will be recruited from the Washingington University Neurofibromatosis-1 (NF1) Patient Registry Initiative (NPRI) and NF Center Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2012-10; Primary Completion 2017-05-08 (Actual); Study Completion 2017-05-08 (Actual)

PRIMARY OUTCOMES:
Brain Tumor | September 1, 2012-February 1, 2014

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly J Johnson, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided